CLINICAL TRIAL: NCT06418126
Title: Prediction of Radiotherapy Efficacy in Patients With Triple-negative Breast Cancer : TNBC-RT2023
Brief Title: Prediction of Radiotherapy Efficacy in Patients With Triple-negative Breast Cancer
Acronym: TNBC-RT2023
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-003
Record Dates: First submitted 2024-04-11; First posted 2024-05-16 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Triple-negative Breast Cancer
Keywords: Radiotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with TNBC breast cancer (Experimental): Patients will be recruited before the start of radiotherapy. A blood sample (20 ml) will be taken before radiotherapy and immediately after the 4th radiotherapy session.
  They will be followed up annually for 5 years after the end of treatment, to determine whether their cancer has recurred.
  Interventions: Biological: blood sampling before radiotherapy; Biological: blood sampling after the fourth radiotherapy session; Other: collection of acute toxicity (radiodermatitis); Other: collection of late toxicity; Other: collection of disease status; Radiation: Radiotherapy - Breast +/- lymph node areas; Radiation: Radiotherapy - Boost operating bed

INTERVENTIONS:
Biological: blood sampling before radiotherapy — A blood sample (20 ml) will be taken prior to radiotherapy
Biological: blood sampling after the fourth radiotherapy session — A blood sample (20 ml) will be taken immediately after the 4th radiotherapy session.
Other: collection of acute toxicity (radiodermatitis) — for the entire duration of radiotherapy
Other: collection of late toxicity — every year for 5 years
Other: collection of disease status — throughout the study
Radiation: Radiotherapy - Breast +/- lymph node areas — 40.05 Gy in 15 fractions of 2.67 Gy, one fraction per week, 5 days per week Or 50 Gy in 25 fractions of 2 Gy, one fraction per week, 5 days per week
Radiation: Radiotherapy - Boost operating bed — 10 Gy in 4 fractions of 2.5 Gy, one fraction per week, 5 days per week Or 16 Gy in 8 fractions of 2 Gy, one fraction per week, 5 days per week

SUMMARY:
Recurrence of triple-negative breast cancer (TNBC) occurs in around 30% of patients within 3 years of treatment. For some TNBC patients, recurrence occurs on average 2.6 years after treatment, while for others recurrence does not occur early. TNBC patients can therefore be divided into two groups: those with early recurrence and those who respond well to treatment.

At present, there are no biomarkers to differentiate these two groups. Some studies suggest that radiation-induced inflammatory cytokines may stimulate the development of new metastases. Gene expression profiling or protein signatures have not been able to define such biomarkers.

The aim of this research protocol is to recruit patients to evaluate if the elevation of the cytokines IL-1β, IL-5 and IL-6 in plasma collected during radiotherapy can be used to predict TNBC patients at high risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

Women with TNBC breast cancer who meet the following criteria:

* Women aged 18 and over;
* Any tumor size (pT stage);
* Regional lymph node pN0 to pN3;
* Patient with pathologically confirmed TNBC (estrogen and progesterone receptor negative and HER2 negative);
* Neo- or adjuvant chemotherapy followed by radiotherapy;
* No evidence of distant metastasis at time of diagnosis;
* Primary tumor removed by conservative surgery with negative margins;
* Patient covered by the French social security system (for French patients).

Exclusion Criteria:

* Distant metastasis at the time of diagnosis;
* Pregnant or breast-feeding women;
* Woman deprived of liberty, under guardianship or trusteeship.
* Patient unable to give consent
* Patient unable to speak French
* Patients unable to undergo regular long-term surveillance.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2030-08-19 (Estimated)

PRIMARY OUTCOMES:
Predictive value of recurrence associated with the appearance of inflammatory cytokines | up to 5 years
  Determine whether TNBC patients who respond poorly to radiotherapy can be identified by the appearance of inflammatory cytokines in the blood during radiotherapy.

SECONDARY OUTCOMES:
To determine whether the increased invasive capacity of TNBC cells incubated with plasma collected during radiotherapy will be associated with recurrence. | up to 5 years
  TNBC cells will be incubated with plasma collected before or during radiotherapy. Boyden chambers will be used to determine the increase in cell invasion.
To determine whether the development of metastases in a mouse model injected with TNBC D2A1 cells pre-incubated with plasma collected during radiotherapy will be associated with recurrence. | up to 5 years
  Number and sizes of metastases to the lungs will be determined after i.v. plasma injection in Balb/c mice.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg europe, Strasbourg, France